CLINICAL TRIAL: NCT04050449
Title: Observational Cohort to Assess Therapeutic Efficacy and Emergence of HIV Drug Resistance Following Initiation of Tenofovir-Lamivudine-Dolutegravir (TLD) for First- or Second-Line ART or With Rifampin-Containing TB Treatment: The Hakim Study
Brief Title: Assess Therapeutic Efficacy and Emergence of HIV Drug Resistance Following Initiation of TLD
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ACTG A5381; UM1AI068636 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Switch to TLD from NNRTI first-line regimen: Participants switching to TLD from a first-line regimen containing a NNRTI. These participants will be divided into two subgroups based upon their HIV-1 RNA level in a sample obtained at entry, before starting TLD. Group 1a will include participants with viremia (HIV-1 RNA >1000 copies/mL at start of TLD) and Group 1b will include participants with suppressed viral load (HIV-1 RNA ≤1000 copies/mL at start of TLD).
- Group 2: Switch to TLD from boosted PI second-line regimen: Participants switching to TLD from a second-line regimen containing a boosted PI. These participants will be divided into two subgroups based upon their HIV-1 RNA level in a sample obtained at entry, before starting TLD. Group 2a will include participants with viremia (HIV-1 RNA >1000 copies/mL at start of TLD) and Group 2b will include participants with suppressed viral load (HIV-1 RNA ≤1000 copies/mL at start of TLD).
- Group 3: Concomitant TLD and RIF-containing TB treatment: Participants initiating concomitant TLD and RIF-containing TB treatment, with an additional daily dose of dolutegravir (DTG) 50mg. For participants already on RIF-containing TB treatment when TLD treatment is started, TLD treatment must be started within 8 weeks (56 days) of the start of RIF-containing TB treatment. Group 1, 2, or 4 participants who start RIF-containing TB treatment after enrollment will have additional evaluations at the start and end of concomitant HIV and TB treatment but will not be co-enrolled in Group 3 (their additional evaluations will, however, be considered when analyzing data from Group 3).
- Group 4: ART-naive initiating TLD therapy: Antiretroviral therapy (ART)-naïve participants initiating therapy with TLD

SUMMARY:
Tenofovir disoproxil fumarate/lamivudine/dolutegravir (TLD) is being used more widely across the world to treat HIV. This is an observational study (a type of study in which participants are observed and certain outcomes are measured). The aim of this study is to observe how successful TLD is at treating HIV, in the following groups of people:

* People switching to TLD, after taking anti-HIV medication that contains a nonnucleoside reverse transcriptase inhibitor (NNRTI) drug (such as Efavirenz or Nevirapine) (Group 1).
* People switching to TLD, after taking anti-HIV medication that contains a boosted protease inhibitor (PI) drug (such as Lopinavir or Atazanavir) (Group 2).
* People taking TLD and receiving medication for TB that includes the drug rifampicin (RIF) (Group 3). These people must be starting one or both of these medications when they enter the study.
* People starting TLD who have not taken anti-HIV medication before (Group 4).

Another goal of this study is to use genetic testing of the virus (HIV) to see how often HIV is resistant to TLD. Genetic testing of the virus is one way to see if the TLD medication is not working to treat a person's HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at a PEPFAR-supported site.
* Documentation of HIV-1 infection acceptable to the local PEPFAR-supported program to allow ART to be initiated or continued.
* Ability and willingness of participant or legal guardian/representative to provide informed consent to participate in the study.
* Expectation that the participant will receive care within the local PEPFAR-supported program and will be able to be followed for study evaluations for at least 6 months and ideally for 36 months.
* Group 1 participants: Receipt of an NNRTI-containing first-line ART regimen from a clinic in a PEPFAR-supported country for at least 6 consecutive calendar months prior to study entry. NOTE: ART treatment gaps are allowed, but treatment gaps should not exceed 14 consecutive days in the 6 calendar months prior to study entry.
* Group 1 participants: HIV-1 RNA >1000 copies/mL obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.
* Group 2 participants: Receipt of a boosted PI-containing second-line ART regimen from a clinic in a PEPFAR-supported country for at least 6 consecutive calendar months prior to study entry. NOTE: ART treatment gaps are allowed, but treatment gaps should not exceed 14 consecutive days in the 6 calendar months prior to study entry.
* Group 2 participants: HIV-1 RNA obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.

  1. If Group 2b reaches its enrollment target of 360 participants, the protocol team will notify sites that the following criteria will be implemented: For Group 2 participants, an HIV-1 RNA >1000 copies/mL will need to be obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry.
  2. If Group 2a reaches its enrollment target of 180 participants, the protocol team will notify sites that the following criteria will be implemented: For Group 2 participants, an HIV-1 RNA ≤1000 copies/mL will need to be obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry.
* Group 4 participants: No current or prior ART treatment. NOTE: Women who received ART regimens only during pregnancy and/or breastfeeding for prevention of mother-to-child transmission but who have not taken any ART drugs for at least 6 calendar months immediately prior to study entry will be allowed.
* For Group 1, 2, and 4 participants, expected initiation of TLD taken once daily within 7 days after study entry. NOTE: Group 1, 2, and 4 participants may not be on, or expected to start, RIF-containing TB treatment at the time of study entry.
* For Group 3 participants already on RIF-containing TB treatment but not on TLD at study entry, expected initiation of TLD taken once daily with an additional daily dose of DTG 50 mg. This must be started within 7 days after study entry AND within 56 days after the start of RIF-containing TB treatment. These participants may be ART-naïve, or may be switching from a first- or second-line ART regimen. NOTE: For ART-naïve participants who start RIF-containing TB treatment first and then start TLD at a later date, screening must occur within 14 days before the intended TLD start date.
* For Group 3 participants not already on RIF-containing TB treatment but already on TLD at study entry, receipt of TLD for at least 6 consecutive calendar months prior to study entry AND expected initiation of RIF-containing TB treatment within 7 days after study entry.
* For Group 3 participants not already on RIF-containing TB treatment or TLD at study entry, expected initiation of TLD and RIF-containing TB treatment within 7 days after study entry. These participants may be ART-naïve, or may be switching from a first- or second-line ART regimen.
* For Group 1 participants, HIV-1 RNA >1000 copies/mL obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.
* For Group 2 participants, HIV-1 RNA obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.

  1. If Group 2b reaches its enrollment target of 360 participants, the protocol team will notify sites that the following criteria will be implemented: For Group 2 participants, an HIV-1 RNA >1000 copies/mL will need to be obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry.
  2. If Group 2a reaches its enrollment target of 180 participants, the protocol team will notify sites that the following criteria will be implemented: For Group 2 participants, an HIV-1 RNA ≤1000 copies/mL will need to be obtained as part of standard of care or with a real-time test within 12 weeks prior to study entry.

Exclusion Criteria:

* Weight ≤30 kg.
* For participants already on ART in Groups 1, 2, and 3, known to have had an ART interruption encompassing the entire 14 day window (≥14 consecutive days) immediately prior to study entry.
* For Group 3, if a participant is already taking TLD at the time of study entry, HIV-1 RNA >1000 copies/mL within the past 9 months while taking TLD with no subsequent HIV-1 RNA ≤1000 copies/mL.
* Prior enrollment in any group in this study.
* For Group 3 participants, already on concomitant TLD and RIF-containing TB treatment prior to study entry.
* For Group 2 participants with HIV-1 RNA >1000 copies/mL from a host country in which treatment guidelines require a genotypic test prior to switching patients on a boosted PI-containing second-line ARV regimen to TLD, 65R RT mutation within 12 weeks prior to study entry.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected adults and adolescents (>30 kg, ≥10 years of age) initiating or switching to TLD and receiving care through a President's Emergency Plan for AIDS Relief (PEPFAR)-supported treatment program.
Sampling Method: Non-Probability Sample
Enrollment: 1339 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving virologic success at 6 months (Groups 1, 2, and 4) | 6 months +/- 3 months after starting TLD
  Proportion of participants on TLD at 6 months achieving virologic success, defined as suppression of plasma HIV-1 RNA to ≤1000 copies/mL. This will be based on the measurement closest to exactly 6 months (i.e., 183 days) after the date of start of TLD, within the window of 6 months ±3 months (specifically 92 to 274 days, inclusive).
Proportion of participants achieving virologic success at end of TLD and RIF-Containing TB Treatment (Group 3) | 4 weeks before to 6 months after end of TLD and RIF-containing TB treatment (expect to end concomitant treatment within 12 months of study entry)
  Proportion of participants achieving virologic success, defined as suppression of plasma HIV-1 RNA to ≤1000 copies/mL at the end of concomitant TLD and RIF-containing TB treatment. This will be the measurement closest to the end of concomitant treatment within the window of 4 weeks (28 days) before the end to 6 months (183 days) after the end, inclusive.

SECONDARY OUTCOMES:
Proportion of participants achieving virologic success | 6 months, 12 months, 24 months, and 36 months after starting TLD
  Based on the FDA Snapshot algorithm modified to use the HIV-1 RNA threshold of 1000 copies/mL (instead of the usual 50 copies/mL) at 6 months, 12 months, 24 months, and 36 months after starting TLD in each of Groups, 1a, 1b, 2a, 2b, and 4; and at the end of concomitant TLD and RIF-containing TB treatment, 12 months, 24 months, and 36 months after starting concomitant TLD and RIF-containing TB treatment in Group 3.
Proportion of participants with low HIV-1 RNA | 12months, 24 months, and 36 months.
  Plasma HIV-1 RNA ≤1000 copies/mL
Time to confirmed virologic failure (VF) | At or after 6 months which is confirmed by the next HIV-1 RNA measurement
  Time to confirmed virologic failure (VF), defined as the time from start of TLD to the first HIV-1 RNA >1000 copies/mL at or after 6 months which is confirmed by the next HIV-1 RNA measurement also being >1000 copies/mL
Time to confirmed virologic failure with a new DTG resistance-associated mutation | From 0 to 36 months
  DTG resistance-associated mutation as detected in population-based sequencing. New is a mutation not present in the last population-based sequence obtained prior to initiating TLD).
Time from start of TLD to TLD discontinuation | From 0 to 36 months
  Time from start of TLD to TLD discontinuation
Time from start of TLD to TLD discontinuation due to toxicity. | From 0 to 36 months
  Time from start of TLD to TLD discontinuation due to toxicity.
Change in quality of life (QoL) | From study start to 6 months
  Change in quality of life (QoL), defined as the difference in the summary scores obtained from the ACTG SF-21 at 6 months from the scores obtained at study entry
Time from start of TLD to first occurrence of a targeted clinical event | From 0 to 36 months
  Time from start of TLD to first occurrence of a targeted clinical event

CONTACTS AND LOCATIONS:
Overall Officials: Cissy Kityo, MBChB; M.Sc.; Ph.D., Study Chair — Joint Clinical Research Centre (JCRC)/Kampala CRS
Locations (14):
- Haiti (2):
  - Les Centres GHESKIO CRS (30022), Port-au-Prince, Bicentaire
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS (31730), Port-au-Prince
- Kenya (3):
  - Moi University Clinical Research Center (MUCRC) CRS (12601), Eldoret
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS (12501), Kericho
  - Kisumu Crs (31460), Kisumu
- Malawi (2):
  - Blantyre CRS (30301), Blantyre
  - Malawi CRS (12001), Lilongwe
- South Africa (5):
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (11101), Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CUR) CRS (8950), Cape Town, West Cape
  - University of Cape Town Lung Institute (UCTLI) CRS (31792), Cape Town, Western Cape
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
- Joint Clinical Research Centre (JCRC)/Kampala CRS (12401), Kampala, Uganda
- Milton Park CRS (30313), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: Related Info — https://actgnetwork.org

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT04050449/Prot_ICF_000.pdf